CLINICAL TRIAL: NCT02376062
Title: Bundled Intervention Integrating Mental Health Service Into Rural Primary Care in Nepal: Implementation Research Study
Brief Title: Bundled Intervention Integrating Mental Health Services in Nepal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Possible (Other)
Collaborators: University of California, San Francisco (Other); Harvard Medical School Center for Global Health Delivery-Dubai (Unknown); National Institute of Mental Health (NIMH) (NIH); Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MHCMEnyaya
Record Dates: First submitted 2014-12-31; First posted 2015-03-03 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Mental Health
Keywords: Continuing Medical Education; Chronic Diseases; Nepal; Implementation Research
MeSH Terms: conditions — Psychological Well-Being; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bundled Intervention (Experimental): * On-site care coordinator and off-site psychiatric supervisors based in Nepal's capital, Kathmandu
  * Weekly case conferences
  * Surveys of clinicians and clinical supervisors in accordance with CME curriculum
  Interventions: Other: Bundled Intervention

INTERVENTIONS:
Other: Bundled Intervention — The authors have designed continuing medical education curriculum to improve clinical capacity and competency about mental health for Nepali Primary Care Providers. Specifically:
  * On-site care coordinator and off-site psychiatric supervisors based in Nepal's capital, Kathmandu
  * Weekly case conferences
  * Surveys of clinicians and clinical supervisors in accordance with CME curriculum

SUMMARY:
Globally, access to mental healthcare is often non-existent in rural, resource-deprived communities despite the pervasive need for services, particularly in post-conflict and post-disaster settings. We are developing and piloting will develop and pilot a culturally appropriate training model for non-specialist providers (NSPs) to deliver high-quality mental health care over a period of 24 months in a primary care hospital in a rural district in Nepal. We will employ a mixed methods framework to evaluate change in skills, knowledge, and attitude in NSP's, identify key mechanisms for continuum of mental healthcare delivery, and efficacy and cost-effectiveness in care delivery through a government hospital, clinics, and a network of community health workers. This integrated approach will introduce a bundled intervention that includes: both an on-site care coordinator and off-site psychiatric supervisors based in Nepal's capital, Kathmandu, weekly case conferences, and surveys of NSP's and clinical supervisors every six months during the study period. To learn about the acceptability, feasibility and challenges in the program we will also conduct Focus Group Discussions among the PCPs. In the last one year of the research in Achham District we have seen increase in knowledge efficacy and skills among the NSPs and also improved mental health care services at Bayalpata Hospital. Our experience in Achham motivated us to develop a similar program for Charikot Primary Health Center in Dolakha District. Outcomes of this study will focus on efficacy of this model to appropriately identify, counsel, and treat patients with depression, psychosis, and post-traumatic stress disorder (PTSD) through an integrated rural mental healthcare delivery intervention as a model for rural healthcare delivery.

ELIGIBILITY:
Inclusion Criteria:

* Primary Care Provider (MBBS-level physician or Health Assistant)
* Current staff at healthcare facility in Achham, Bajura, or Doti Districts.

Exclusion Criteria:

* N/A

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2016-02-06 (Actual); Primary Completion 2019-07-30 (Estimated); Study Completion 2019-07-30 (Estimated)

PRIMARY OUTCOMES:
Changes in knowledge, attitudes, practices, and self-efficacy of Primary Care Providers | 3 years
  To measure retention of knowledge, and change in attitudes, practices, and self-efficacy among primary care providers who take part in the integrated mental health care delivery intervention. The primary outcome will be reported as change in scores for all pre-and post-tests will be scored with a total score of 100 on each module. Self-efficacy will be assessed on a Likert Scale. Change in knowledge and self-efficacy before and after the intervention will be compared with wilcoxon rank sum tests, assuming lack of normal distribution and given the small sample size. Trainee's rating of the module will be on a Likert scale from 1-5 and these will be presented as means with standard deviation.
Longitudinal clinical outcomes for patients with depression, post-traumatic stress disorder, and patient self-reported medication adherence | 3 years
  To analyze the longitudinal clinical outcomes related to a decrease in acute symptoms as measured by PHQ-9 and PCL, regular adherence to medication and counseling as appropriate. The primary outcome will be reported as the difference in means of the PHQ-9 scores (depression) or PCL scores (post-traumatic stress disorder) before and after the length of the intervention. For patients who are lost of follow-up, the last observation will be carried forward. For patient self-reported medication adherence, the primary outcome will be patient self reported rates of medication adherence, based on a "Yes" response to the question "Have you been able to take your medications as prescribed almost all the time?".
Cost assessment of bundled intervention | 3 years
  To assess the costs and scalability of the bundled intervention through mixed quantitative and qualitative methods. We will include the following expenses aggregated to per patient per year psychotropic medications, time effort for PCPs, psychosocial counselors, consultant psychiatrist and nurses, and laboratory and other diagnostic tools.

CONTACTS AND LOCATIONS:
Overall Officials: David Citrin, PhD, MPH, Study Director — Possible
Locations (2):
- Nepal (2):
  - Bayalpata Hospital, Sanfebagar, Achham
  - Charikot Primary Health Center, Bhimeshwor, Dolakha

REFERENCES:
- See also: Possible — http://possiblehealth.org
- See also: Healthcare Systems Design Group — http://hsdg.partners.org/